CLINICAL TRIAL: NCT01479478
Title: Oral Probiotic Supplementation and Group B Streptococcus Rectovaginal Colonization in Pregnant Women: a Randomized Double-blind Placebo-controlled Trial.
Brief Title: Effects of Oral Probiotic Supplementation on Group B Strep (GBS) Rectovaginal Colonization in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Natali Aziz, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18840
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Infection; Pregnancy
MeSH Terms: conditions — Infections | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic dietary supplement (Active Comparator): Probiotic dietary supplement one capsule once per day until delivery.
  Interventions: Dietary Supplement: Probiotic dietary supplement
- Placebo (Placebo Comparator): Placebo capsule, one daily until delivery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — One placebo capsule daily.
  Other Names: Sugar pill
  Arms: Placebo
Dietary Supplement: Probiotic dietary supplement — Dietary Supplement: Lactobacillus rhamnosus GR-1, Lactobacillus reuteri RC -14
  Other Names: Other Names:; Jarrow's fem-dophilus
  Arms: Probiotic dietary supplement

SUMMARY:
The investigators wish to determine if oral probiotic supplementation during the second half of pregnancy decreases maternal GBS recto-vaginal colonization at 35-37 weeks' gestational age, thereby decreasing need for maternal antibiotic administration at time of labor. The importance of this study is that it may offer a safer alternative to antibiotic treatment of group B Streptococcus (GBS) colonized pregnant women.

DETAILED DESCRIPTION:
1. Screening: All pregnant women prior to 28 weeks gestational age. Patients who choose to enroll and who will not deliver at Lucile Packard Childrens Hospital at Stanford will sign release of medical information forms for study personnel to access pregnancy outcomes. Patients receiving obstetric care at any of the satellite research sites in Santa Cruz will also be offered enrollment in the study.
2. Women will continue regular and routine obstetric care and clinic visits.
3. Placebo vs probiotic daily regimen: We plan to begin administration of product and placebo at 20 weeks gestation, and no later than 28 weeks gestation until delivery. Once a women is enrolled in the study, she will be randomized to either the placebo or the probiotic group.
4. At the time of randomization, the patient will receive her month supply of 30 capsules; The allocation arm will be double-blinded.
5. The investigators will schedule the women for routine monthly obstetric visits (more often if clinically required) during which time they will also meet with one of the investigators. The investigator at each monthly visit will provide an additional monthly allotment of 30 capsules. The capsule bottle from the previous cycle will be collected and dated if there are capsules remaining in the bottle. Remaining capsules will be counted and refrigerated for future use.
6. The investigators will collect history data including safety data per the questionnaire and will document compliance with the study.
7. GBS recto-vaginal screening: The investigators will enroll the women in the study and we will perform the standard GBS colonization screening (using standard GBS recto-vaginal cultures) at 36 weeks.
8. Additionally, subjects may opt to have serial vaginal swabs collected to assess potential beneficial effects of probiotics on the vaginal microbiota and bacterial vaginosis (BV) status. Vaginal swabs will be collected (either by study personnel or self-collected by the study participant). Swabs will be inserted 1-2 inches into the vaginal introitus and spun for 20 seconds and then withdrawn. Swabs will be collected at the following time points: prior to probiotic/placebo initiation, every 1-4 weeks from time of enrollment to time of delivery, and postpartum serially up to 12 months. These swabs will be stored at -20 degrees Celsius or colder for additional microbiologic analyses.
9. Additionally, placental tissue may be collected at time of delivery for possible future microbiome and/or other analyses.
10. Women who suffer a premature rupture of the membranes, deliver before 36 weeks gestation, or go into labor before the GBS culture result is available, will receive the standard GBS antibiotic prophylaxis.
11. Labor: The patient will receive standard delivery and newborn care. Patients with a positive GBS culture will be treated with standard antibiotics in labor.
12. Postpartum and neonatal care: The patient will receive routine postpartum care per the obstetric team. Data regarding her postpartum course and neonatal outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 20-28 weeks gestation.
2. 18 years of age or older.
3. Singleton gestation.

Exclusion Criteria:

1. Preexisting morbidity: Immunocompromised status (HIV +; malignancy; history of organ transplant; chronic steroid therapy; autoimmune disease requiring treatment during pregnancy, and other immunocompromised states); Type 1 diabetes and type 2 diabetes;congenital cardiac disease and cardiac valvular disease requiring antibiotic prophylaxis during procedure/labor; pulmonary disease (except mild asthma); renal disease; chronic hepatic disease (Hepatitis B, C); inflammatory bowel disease (Crohn's disease or ulcerative colitis); stomach or duodenal ulcer; bowel resection, gastric bypass, and chronic indwelling venous, bladder, or gastric catheter.
2. Multi-fetal gestation.
3. Use of probiotics preparations in the 3 months prior to beginning of the study treatment or use of any additional probiotics preparations (other than study treatment) at any time during the study period (including over the counter food supplements such as Activia, BioK, other oral or vaginal probiotics products (BUT not including other common forms of yogurt).
4. Chronic (daily) use of broad spectrum antibiotics.
5. History of infant with GBS sepsis.
6. Intrauterine Growth Restriction (IUGR), Fetal Anomalies-major diagnosed at time of second trimester anatomy ultrasound
7. Anticipated delivery <35 wks for maternal/fetal indication
8. Placenta previa or accreta (with anticipated delivery prior to 35 weeks)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 251 (Actual)
Dates: Start 2011-11; Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natali Aziz, MD, Principal Investigator — Stanford University School of Medicine/Lucile Packard Children's Hospital
Locations (3):
- United States (3):
  - Aptos Women's Health Center, Aptos, California
  - Dominican Hospital, Santa Cruz, California
  - Stanford University School of Medicine/Lucile Packard Children's Hospital, Stanford, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only expecting mothers were enrolled in this study. Neonatal data were collected from respective pregnancies, however, the neonates were not considered to be enrolled in this study.
Period: Overall Study
Arm/Group | Probiotic Dietary Supplement | Placebo
Started | 125 | 126
Completed | 125 | 126
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic Dietary Supplement | Placebo | Total
Number analyzed (Participants) | 125 | 126 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (5.7) | 31.9 (5.3) | 31.7 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 126 | 251
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic white | 66 | 71 | 137
  Non-Hispanic other | 21 | 22 | 43
  Hispanic | 32 | 26 | 58
  Unknown | 6 | 7 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 125 | 126 | 251
Pre-pregnancy Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (6.5) | 26.0 (7.5) | 26.1 (7)

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Positive Group B Streptococcus Rectovaginal Colonization Status at 35- 37 Weeks' Gestational Age
Description: Gestational age is given in a format of full weeks.
Time Frame: 35 to 37 weeks gestational age
Population: Participants with available data were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 108 | 117
Participants | 20 | 23
Statistical Analysis 1: Comparison: Probiotic Dietary Supplement vs Placebo; Test type: Superiority; p = 0.87, Cochran-Mantel-Haenszel

2. Secondary Outcome: Count of Participants With Urinary Tract Infection
Time Frame: From enrollment up to delivery hospitalization (up to 42 weeks gestation)
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 118 | 123
Participants | 8 | 9

3. Secondary Outcome: Count of Participants With Intrapartum Chorioamnionitis
Description: Intrapartum chorioamnionitis is maternal temperature above 38.0 degrees Celsius and one or more of the following findings: fetal tachycardia; maternal tachycardia; uterine tenderness; purulent or malodorous amniotic fluid, or elevated maternal white blood cell count.
Time Frame: From time of labor onset until delivery (up to 42 weeks of gestation)
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 118 | 121
Participants | 5 | 4

4. Secondary Outcome: Count of Participants With Endometritis
Description: Endometritis is a uterine (myometrial) infection.
Time Frame: From time of delivery up to 6 weeks postpartum
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 116 | 119
Participants | 0 | 2

5. Secondary Outcome: Count of Participants With Cellulitis
Description: Cellulitis is a bacterial skin infection.
Time Frame: From time of delivery up to 6 weeks postpartum
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 118 | 123
Participants | 0 | 0

6. Secondary Outcome: Count of Participants With Bacteremia
Description: Bacteremia is defined as presence of bacteria in the blood.
Time Frame: From time of labor onset up to 6 weeks postpartum
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 116 | 119
Participants | 0 | 0

7. Secondary Outcome: Count of Participants With Sepsis
Description: Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated response of the body to an infection.
Time Frame: From labor onset up to 6 weeks postpartum
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 116 | 119
Participants | 0 | 0

8. Secondary Outcome: Count of Participants With Other Infectious Morbidity
Description: Other infectious morbidity included maternal mastitis or pneumonia.
Time Frame: From time of labor onset up to 6 weeks postpartum
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 116 | 119
Participants | 0 | 0

9. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age at delivery is presented as weeks.
Time Frame: At time of delivery (up to 42 weeks of gestation)
Population: Participants with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 117 | 121
weeks | 39.6 [39.0 to 40.6] | 39.4 [38.7 to 40.3]

10. Secondary Outcome: Apgar Score at 1 and 5 Minutes Following Delivery
Description: Apgar score is a measure to quickly assess the neonatal health status from time of delivery. Score ranges from 0-10. Lower scores correspond to worse health state; neonates with scores below 5 are considered to have poor prognosis.
Time Frame: At time of delivery (up to 42 weeks of gestation)
Population: Participants with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 113 | 119
units on a scale
  At 1 minute | 8 [7 to 9] | 8 [8 to 9]
  At 5 minutes | 9 [9 to 9] | 9 [9 to 9]

11. Secondary Outcome: Neonatal Bilirubin Level
Time Frame: Up to 14 days following delivery
Population: Participants with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 104 | 94
mg/dL | 6.4 [5.1 to 9.6] | 6.5 [4.9 to 9.4]

12. Secondary Outcome: Neonatal C-reactive Protein Level
Description: Maximum neonatal C-reactive protein level
Time Frame: Up to 14 days following delivery
Population: Participants with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 23 | 18
mg/L | 1.6 [0.3 to 4.1] | 1.2 [0.4 to 2.9]

13. Secondary Outcome: Count of Neonates Requiring a "Rule-out Sepsis Evaluation"
Description: Outcome was based on performance of neonatal blood culture.
Time Frame: Up to 14 days following delivery
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 115 | 121
Participants | 9 | 4

14. Secondary Outcome: Count of Neonates With Sepsis
Time Frame: Up to 14 days following delivery
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 115 | 121
Participants | 4 | 1

15. Secondary Outcome: Count of Neonates With Pneumonia
Time Frame: Up to 14 days following delivery
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 115 | 121
Participants | 0 | 0

16. Secondary Outcome: Count of Neonates With Meningitis
Time Frame: Up to 14 days following delivery
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 115 | 121
Participants | 0 | 0

17. Secondary Outcome: Count of Neonates With Intensive-care Unit Admission
Time Frame: Up to 14 days following delivery
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 115 | 121
Participants | 12 | 7

18. Secondary Outcome: Length of Neonatal Hospital Stay
Time Frame: Up to 14 days following delivery
Population: Participants with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Probiotic Dietary Supplement | Placebo
Number analyzed (Participants) | 113 | 116
days | 2 [2 to 3] | 2 [2 to 2.5]

ADVERSE EVENTS:
Time Frame: From enrollment up to 6 weeks following delivery.
Arm/Group | Probiotic Dietary Supplement | Placebo
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/126
Serious Adverse Events (participants affected / at risk) | 1/125 | 0/126
Other Adverse Events (participants affected / at risk) | 0/125 | 0/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Probiotic Dietary Supplement (N=125) | Placebo (N=126)
Any other anticipated or unanticipated life-threatening event:intra-uterine fetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2013-11-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT01479478/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT01479478/SAP_001.pdf